# COVER SHEET

Informed consent document

Study Identifier: NCT04202757

Brief Title: Intravenous Plasma Treatment for Parkinson's Disease (yFFP)
Official title: Intravenous young Fresh Frozen Plasma (yFFP) Investigational Treatment for
Parkinson's Disease

Last document revision: Jan. 14, 2020 IRB approval date: Feb. 7, 2020 IRB: Institute of Regenerative and Cellular Medicine

# **Informed Consent**

**Study:** Intravenous young Fresh Frozen Plasma (yFFP) Investigational Treatment for Parkinson's Disease – Randomized Controlled Study

Study Number: YP102018v3

**Study Presenter:** Dr. Dian Ginsberg, MD

**Co-Investigators:** Dr. Igor Cherches, MD

Dr. Eddie Patton, MD

Study Site: The Neurology Center

6655 Travis St Suite 600 Houston, TX 77030 (713) 795-0074

### Introduction

Please read this form carefully. It is a patient consent form for you to participate in an experimental, clinical trial, and to authorize limited disclosure of your health information. If you agree to take part in this study, you need to sign this form. Your signature means you have been told about, and understand, the study and what the risks are. Your signature on this form also means you wish to take part in this study.

We invite you to take part in a research study: Intravenous young Fresh Frozen Plasma (yFFP) Investigational Treatment for Parkinson's disease – Randomized Controlled Study, which seeks to identify a more effective means of treating those conditions. Taking part in this study is entirely voluntary. We urge you discuss any questions about this study with our staff members. Talk to your family and friends about it and take your time to make your decision. If you decide to participate you must sign this form to show that you want to take part.

### Section 1. Purpose of the Study

The purpose of this study is to inquire whether infusions of plasma collected from 18- to 25-year-old volunteer donors (yFFP) improves or slows the progression of cognitive, mood and/or motor impairment and rate markers of the disease.

As neurodegenerative diseases progress, there are major changes throughout the body and brain. These changes are transmitted in the body via the circulatory system between organs, tissues and cells. Recent findings have shown that infusions of yFFP can have beneficial effects on cognitive functions. This suggests that the circulating components of yFFP can improve cognitive and disease-relevant symptoms.

The long-established safety of blood plasma infusions allows the investigators to test whether infusions of young plasma can ease the neurological symptoms in human subjects with neurodegenerative diseases. This study will address a well known neurological disorder for which there are few effective treatments and an urgent need to find an efficacious management that could help prevent, or at least slow down the progress of these major public health problems.

Approximately twenty people will take part in this study in Houston.

#### Section 2. Procedures

This study is a prospective, randomized double-blind, placebo-controlled trial, designed to evaluate the efficacy of intravenous young Fresh Frozen Plasma at 12.5 ml/kg in each of two doses, one day apart (25 ml/kg total).

Placebo group patients receive an infusion n of 0.9% Sodium Chloride with Vitamin B2 as riboflavin 5-phosphate sodium solution added for the color match, at a volume rate equal to that of yFFP 12.5 ml/kg in each of two doses, one day apart.

Consecutive patients are randomly (blind) assigned to one of the two treatment study groups, labeled 'yFFP' or 'Saline' group.

# Section 3. Time Duration of the Procedures and Study

For the time frame, study day 0 is defined as the day of randomization, and a screening visit is scheduled maximally two weeks prior to first infusion; patients then receive blinded infusions on days 1 and 2. The average infusion duration for a participant of 75 kg to 90 kg body weight is about 1.5 to 2 hours.

Physician assessments, caregiver surveys and blood tests will be completed at 4-weeks, 12-weeks and 24 weeks, to explore the duration of yFFP - and unspecific treatment effects.

The end of the study will be the last participant's final contact at 6 months

#### Section 4. Discomforts and Risks

Although blood plasma has been in continuous use since the 1920s and 10,000 units are administered each day in the United States, adverse risks are rare and will vary from person to person, while on the study, you are at risk for the following side effects, listed below.

Drugs such as Benadryl may be given to make some of the side effects, if present, less uncomfortable.

The infusion rate for each participant will start slowly at 2 ml per minute for the first fifteen minutes to confirm if the yFFP is well tolerated before increasing to the standardized rate of 15 ml per minute.

#### Contraindications include:

Absolute contraindications to the use of yFFP are documented intolerance to plasma or its components or congenital deficiency of immunoglobulin A (IgA) in the presence of anti-IgA antibodies. Relative contraindications are heart failure or pulmonary edema.

#### Additional Cautions:

Patients should avoid citrus and highly acidic fruits (example: strawberries, blueberries, loganberries, cranberries, currants, gooseberries, pineapple etc.) before and for a day after their last infusion, as patient may experience a reaction due to citrate overload.

yFFP can cause adverse reactions:

- Chills, headache, fever, vomiting, allergic reactions, nausea, arthralgia, low blood pressure and mild back pain, which may occur occasionally.
- Increase in serum creatinine level and/or acute renal failure have been observed.
- Very rarely, thromboembolic reactions, such as myocardial infarction, stroke, pulmonary embolism, and deep vein thromboses have occurred.

Details of further spontaneously reported adverse reactions include the following:

- Cardiac disorders: angina pectoris (very rare)
- General disorders and administrations site conditions: rigors (very rare)
- Immune system disorders: anaphylactoid shock (very rare), hypersensitivity (very rare)
- Investigations: blood pressure decreased (very rare)
- Musculoskeletal and connective tissue disorders: back pain (very rare)
- Respiratory, thoracic and mediastinal disorders: dyspnea NOS (very rare); or
- Vascular disorders: shock (very rare).

If you are in the treatment group that receives placebo (inactive substance) your symptoms or condition may worsen or not improve.

### Other Possible Risks Associated with Participating in This Study:

The risks of drawing blood or infusing yFFP include temporary discomfort from the needle stick, bruising, bleeding, and rarely, infection.

#### **Current Standard of Care**

From the national Parkinson's Foundation:

"There is no standard treatment for Parkinson's disease (PD). Treatment for each person with Parkinson's is based on his or her symptoms. Treatments include medication and surgical therapy. Other treatments include lifestyle modifications, like getting more rest and exercise. There are many medications available to treat the Parkinson's symptoms, although none yet that reverse the effects of the disease.

#### Section 5. Potential Benefits

Infusions of yFFP have been shown to counteract the biological processes underlying neurodegeneration. This study has been initiated to determine the extent and duration of neuro-regeneration resulting from two measured infusions of yFFP. Participating patients are expected to realize improvements in motor, cognitive, mood and other non-motor symptoms, however, individual responses will vary and there is no guarantee that you will benefit from being in this research.

The results of this research will be used to guide the future treatment of patients with the same or similar neurodegenerative disease.

### Section 6. Statement of Confidentiality

A description of this study will be available on http:///www.YoungPlasmaStudy.com This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search the web site at any time.

#### 6a. Privacy and confidentiality measures

Your research records that are reviewed, stored, and analyzed will be kept in a secured area and will be labeled with a code number for privacy purposes.

Your code number will be linked to your name, social security number, address, phone number, and date of birth. The list that matches your name with the code number will be kept in a locked file.

In the event of any publication or presentation resulting from the research, no personally identifiable information will be shared.

We will keep your participation in this research study publically confidential to the extent permitted by law. However, it is possible that the following people/groups may inspect and copy records pertaining to this research.

- The U.S. Food and Drug Administration
- The infusion provider's Institutional Review Board
- The National Institutes of Health
- Texas Medical Board

Some of these records inspected and/or copied by the aforementioned people/groups could contain information that personally identifies you. Reasonable efforts will be made to keep the personal information in your research record private and confidential, but absolute confidentiality cannot be guaranteed.

To participate in this research, you must allow the study team to use your health information. If you do not want us to use your protected health information, you may not participate in this study.

People usually have a right to access their medical records. However, due to the fact that this is a blind study, while the research is in progress, you may not be allowed to see or copy certain information that is related to this research study. This is only for the period of the research. You will be allowed to see that information when the entire research project is complete.

Your permission for the use, retention, and sharing of your identifiable health information will expire upon completion of the research study. Any research information in your medical record will be kept indefinitely.

If you choose to participate, you are free to withdraw your permission for the use and sharing of your health information at any time. You must do this in writing.

If you withdraw your permission:

- We will no longer use or share medical information about you for this research study, except when the law allows us to do so.
- We are unable to take back anything we have already done or any information we have already shared with your permission.
- We may continue using and sharing the information obtained prior to your withdrawal if it is necessary for the soundness of the overall research.
- We will keep our records of the care that we provided to you as long as the law requires.

#### Section 7. Costs for Participation

#### 7a. Costs:

There is no cost to participate. Incidental costs to the participant for parking will be reimbursed at the time that they are incurred.

### 7b. Treatment and compensation for injury:

Every effort to prevent injury as a result of your participation will be taken. It is possible, however, that you could develop complications or injuries as a result of participating in this research study. In the event of injury resulting from this research, medical treatment is available, but will be provided at the usual charge. It is the policy of this institution to provide neither financial compensation nor free medical treatment for research-related injury.

### **Section 8.** Compensation for Participation

You will not receive any compensation for being in this research study.

### Section 9. Research Funding

Golden Genesis, Inc., dba NuPlasma is involved in the research through the provision of intravenous solutions (including yFFP) and study support staffing. RTCD is providing sponsorship funding.

## Section 10. Voluntary Participation

Taking part in this research study is voluntary. If you choose to take part in this research, your major responsibilities will include providing your health history, having blood tests taken, undergoing periodic examinations and assessments and undergoing infusions. You do not have to participate in this research. If you choose to take part, you have the right to stop at any time. If you decide not to participate or if you decide to stop taking part in the research at a later date, there will be no penalty or loss of benefits to which you are otherwise entitled.

Your investigator may take you out of the research study without your permission. If your participation in the research ends early, you may be asked to visit the investigator for a final visit.

If you will be participating in another clinical trial or study while in this research, you should discuss the procedures and/or treatments with your physician or the investigators. This precaution is intended to protect you from possible side effects from interactions of research drugs, treatments or testing.

During the course of the research you will be provided with any significant new findings that may affect your willingness to continue participating in this research.

#### Section 11. Contact Information for Questions or Concerns

You have the right to ask any questions you may have about this research. If you have questions, complaints or concerns or believe you may have developed an injury related to this research, contact the Co-Investigators or Trial Manager at **The Neurology Center (713) 795-0074** 

If you have questions regarding your rights as a research participant or you have concerns or general questions about the research, or about your privacy and the use of your personal health information, contact the Co-Investigators or Trial Manager at **The Neurology Center** (713) 795-0074.

If you wish to contact an impartial third party not associated with this study, you may contact a representative of the ethical review board: **JP Faber of the Institute of Regenerative and Cellular Medicine**: (786) 271-2157.

### Signature and Consent/Permission to be in the Research

Before making the decision regarding enrollment in this research you should have:

- Discussed this study with an investigator,
- Reviewed the information in this form, and
- Had the opportunity to ask any questions you may have.

Your signature below means that you have received this information, have asked the questions you currently have about the research and those questions have been answered. You will receive a copy of the signed and dated form to keep for future reference.

| take part in this research. | rm, you inc | iicate tha | at you are voluntarily choosing to |
|---|---|---|---|
| Signature of Participant | Date | <br>Time | Printed Name |
| Participant's Legally Authorized R<br>Authorized Representative is required<br>By signing below, you indicate that yo<br>this research. | for people | e unable | to give consent for themselves |
| Signature of Participant's Legally | <br>Date | Time | Printed Name |

| Witnes | ss to Pat | <u>ient o</u> | r Leg | <u>ıally A</u> ı | <u>uthoriz</u> | <u>ed Re</u> | pres | <u>senta</u> | tive S | <u>Signat</u> | <u>ure</u> : Your | signa | ature |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| below | means | that | you | have | confir | med | the | rese | arch | was | explained | to | the |
| | oant/partio<br>een ansv | • | • | esentati | ve and | any o | ques | tions | he/sh | e has | about the | rese | arch |
| Witne | ss to Pat | ient Si | gnatu | ıre | | Date | . <u> </u> | ime | ——Print | ted Na | ame | | |